CLINICAL TRIAL: NCT00655304
Title: The Effect of Prometheus (R) Liver Support Dialysis on Intracranial Pressure, Cerebral Oxidative Metabolism and Hemodynamics in Patients With Acute Liver Failure
Brief Title: The Effect of Prometheus (R) Liver Support Dialysis on Cerebral Metabolism in Acute Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Peter Nissen Bjerring, MD, Department of Hepatology, Rigshospitelet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALFPROM-001; H-KF-2007-0006
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Acute Liver Failure; Hepatic Encephalopathy; Intracranial Hypertension
MeSH Terms: conditions — Liver Failure, Acute; Hepatic Encephalopathy; Intracranial Hypertension | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treatment with 6-8 hours of Prometheus (R) liver support dialysis
  Interventions: Device: Prometheus (R) liver support dialysis
- 2 (Active Comparator): Treatment with 6-8 hours of CVVHDF
  Interventions: Device: CVVHDF (Continuously Veno-Venous Hemodiafiltration)

INTERVENTIONS:
Device: Prometheus (R) liver support dialysis — 6-8 hours of dialysis
  Arms: 1
Device: CVVHDF (Continuously Veno-Venous Hemodiafiltration) — 6-8 hours of dialysis with the CVVHDF system PrismaFlex offered by Gambro (Sweden).
  Arms: 2

SUMMARY:
The main objective of this study is to investigate the effect of Prometheus liver support dialysis on intracranial pressure, cerebral metabolism and circulation in patients with acute liver failure.

DETAILED DESCRIPTION:
Acute liver failure (ALF) is a highly mortal medical condition often complicated by multiorgan failure. Apart from severe coagulopathy ALF is characterized by onset of hepatic encephalopathy and in many cases intracranial hypertension (ICH) with the risk of cerebral incarceration. The pathogenesis behind ICH is incompletely understood and the therapeutic options are limited. Prometheus (R) liver support dialysis offers a system that apart from regular high-flux hemodialysis to a certain extent is able of removing albumin-bound substances from the patient - a feature that theoretically could benefit patients with ALF.

In this study we intend to investigate the effect of 6-8 hours of Prometheus (R) liver support dialysis on cerebral metabolism, ICH and cerebral bloodflow (CBF) in patients with ALF. The study is designed as a open, prospective and randomized study, where a control-group treated with 6-8 hours of continuously veno-venous hemodiafiltration (CVVHDF) and standard medical treatment (SMT) is compared to the intervention group treated with Prometheus (R) liver support dialysis and SMT. The study is designed as a cross-over study so that included patients will be treated in both groups in a randomized order.

The primary end-points are treatment effect on intracranial pressure, CBF and cerebral oxidative metabolism (lactate/pyruvate-ratio). We use a intracranial monitoring system from Integra/Camino (R) (United States) in combination with CMA microdialysis system and bedside analyzer (CMA-600) (Stockholm, Sweden).

ELIGIBILITY:
Inclusion Criteria:

* acute liver failure
* and grade II-IV encephalopathy
* and persistent raised arterial ammonia-concentration above 150 micromol/L
* and informed consent from closest relative and general practitioner

Exclusion Criteria:

* withdrawal of informed consent
* severe untreated infection
* active bleeding within 48 hours
* suspicion of malignant liver disease
* severe heart insufficiency or middle artery pressure below 60 mmHg in spite of vasoactive therapy
* pregnant or lactating women
* disseminated intravascular coagulation
* clinical suspicion of cerebral damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
treatment effect on cerebral oxidative metabolism (lactate/pyruvate-ratio) | 24 hours

SECONDARY OUTCOMES:
treatment effect on intracranial pressure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Bjerring, MD, Principal Investigator — Department of Hepatology, Rigshospitalet
Locations (1):
- The liverfailure unit, Department of hepatology, Rigshospitalet, Copenhagen, Denmark